CLINICAL TRIAL: NCT04596852
Title: Protocol Validation of Dynamometric Measurement of Passive Inter-segmental Stiffness and Spasticity in Children With Cerebral Palsy: (DYNA_PC)
Brief Title: Protocol Validation of Dynamometric Measurement of Passive Inter-segmental Stiffness and Spasticity in Children With Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ellen Poidatz (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Dyna_PC
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Masking Description: The order of participation of evaluators is random.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy children (Experimental)
  Interventions: Device: Assessment of the reliability of a protocol characterizing intersegmental hyper-resistance to passive stretch
- Children with cerebral palsy (Experimental)
  Interventions: Device: Assessment of the reliability of a protocol characterizing intersegmental hyper-resistance to passive stretch

INTERVENTIONS:
Device: Assessment of the reliability of a protocol characterizing intersegmental hyper-resistance to passive stretch — Passive solicitations of the main joints of the lower limb, of healthy children and children with cerebral palsy, are realized by two evaluators with a handheld dynamometer.
  Repeated measures are performed to assess intra and inter-reliability.

SUMMARY:
Cerebral palsy (CP) refers to a group of movement and posture disorders responsible for activity limitation due to brain damage that occurs during fetal development or during the first year of a child's life.

Given the multitude of treatment options available, the choice of treatment is a key determinant that greatly influences the potential for improvement in motor function. This choice is based in particular on a diagnosis resulting from the comparison of a Clinical Gait Analysis (CGA) and a clinical examination, carried out by a practitioner, aimed at evaluating as accurately as possible the deficiencies present in children with CP.

During the latter examination, passive inter-segmental stiffness and spasticity, both limiting factors in the mobility of the child with CP, are assessed. However, there are significant uncertainties in these measurements, which depend, among other things, on the examiner's feelings. The enrichment of this clinical assessment therefore requires the introduction of quantitative and objective measures. Portable dynamometers are increasingly used to measure the resistance of a joint during passive solicitations.

Thus, both passive inter-segmental stiffness and spasticity can be characterized using instrumental methods. However, in the majority of studies proposed in the literature, the biomechanical computational model used is not unified with that of the CGA, thus altering the approximation of the parameters measured on the table with those estimated during gait. However, in order to evaluate the extent to which these phenomena occur during gait, it is important to follow the same biomechanical calculation procedure.

Thus, our team proposes a new dynamometric measurement protocol for passive inter-segmental stiffness and spasticity adapted to the PC child. Nevertheless, in order to guarantee the reliability of the measurements, manual dynamometric solicitation methods must follow standardized protocols, and their psychometric properties must be defined before they can be used in clinical practice. This is why we wish to study the reliability of this new solution for dynamometric quantification of passive inter-segmental stiffness and spasticity in children with CP.

ELIGIBILITY:
The inclusion criteria for PC children are :

* A clinical diagnosis of CP noted in the medical record
* An age between 7 and 18 years old
* Levels I to III for the Global Motor Function Classification System (GMFCS)
* Ability to cooperate, understand and follow simple instructions
* Patient affiliated to the French social security system
* Voluntary patient whose parents have given their consent to participate

The inclusion criteria for healthy children are :

* An age between 7 and 18 years old
* Ability to cooperate, understand and follow simple instructions
* Patient affiliated to the French social security system
* Voluntary patient whose parents have given their consent to participate

Exclusion Criteria:

* Medical decision for any reason
* Child or parent decision for any reason
* Inability to cooperate, to understand and to follow instructions
* Surgery or botulinum toxin injection within 6 months prior to the start of the study.
* A diagnosis of a form of dystonia.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 85 (Estimated)
Dates: Start 2020-11-02 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Passive Stiffness Index | 2 years
  A stiffness index representing the evolution of the resistance to passive stretch as a function of the angular amplitude.
  A higher score means that the joint is stiffer.
Model deviation | 2 years
  The root mean square deviation between the passive moment predicted by a passive stiffness model, defined at low velocity, and the passive moment measured at high velocity.
  A higher score means that the subject's spasticity is more important.

SECONDARY OUTCOMES:
Electromyography Activity | 2 years
  Electromyography activity during passive solicitations
Joint Kinematics | 2 years
  Joint kinematics during passive solicitations

CONTACTS AND LOCATIONS:
Overall Officials: Eric Desailly, PhD, Principal Investigator — Fondation Ellen Poidatz
Locations (1):
- Fondation Ellen Poidatz, Saint-Fargeau-Ponthierry, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website of the EllenPoidatz Foundation (See Research and Innovation) — https://www.fondationpoidatz.com/